CLINICAL TRIAL: NCT01956136
Title: Efficacy and Neural Basis of Music-based Neurological Rehabilitation for Traumatic Brain Injury
Acronym: MUBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other); Hospital District of Helsinki and Uusimaa (Other); University of Jyvaskyla (Other); Åbo Akademi University (Other); University of Barcelona (Other); University of Virginia (Other); Validia Rehabilitation Helsinki (Unknown)
Responsible Party: Principal Investigator, Teppo Sarkamo, Researcher, PhD, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 141106
Record Dates: First submitted 2013-09-12; First posted 2013-10-08 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Traumatic Brain Injury (TBI)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): The patients receive 10 weeks of Music-based Neurological Rehabilitation (MBNR) and Standard Care (SC) followed by 10 weeks of SC only.
  Interventions: Behavioral: Music-based Neurological Rehabilitation (MBNR); Other: Standard Care (SC)
- Arm 2 (Experimental): The patients receive 10 weeks of Standard Care (SC) only followed by 10 weeks of Music-based Neurological Rehabilitation (MBNR) and SC.
  Interventions: Behavioral: Music-based Neurological Rehabilitation (MBNR); Other: Standard Care (SC)

INTERVENTIONS:
Behavioral: Music-based Neurological Rehabilitation (MBNR) — Music-based Neurological Rehabilitation (MBNR) will involve 10 weeks of individual training (30 sessions, 1 hour per session, 3 days per week) given by a trained music therapist. The MBNR protocol utilizes structured cognitive-motor training with drums (drum set, djembe drums) and creative musical expression (music playing, song writing) with piano that are geared towards engaging and training attention, executive functions, working memory, and upper-extremity functions and for enhancing emotional self-expression, adjustment, and mood after TBI.
Other: Standard Care (SC) — Standard Care (SC) consists of other types of conventional rehabilitation (physical therapy, occupational therapy, speech therapy, and/or neuropsychological rehabilitation) and medical care for TBI that the patients receive in Finnish private or public health care.

SUMMARY:
Traumatic brain injury (TBI) is one of the leading causes of serious, life-long disability among adolescents and young adults. Especially the cognitive, emotional, and motors deficits caused by TBI often impair everyday psychosocial functioning, quality of life and ability to work. The purpose of the study is to determine the long-term effect of music-based rehabilitation on cognitive, motor, emotional, and social recovery after TBI in adolescents and young adults, and to study the neural mechanisms that underlie behavioural recovery and the efficacy of music.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is one of the leading causes of serious, life-long disability among adolescents and young adults. Especially the cognitive, emotional, and motors deficits caused by TBI often impair everyday psychosocial functioning, quality of life (QoL) and ability to work dramatically, thereby bringing about a lot of suffering and burden to the patients and their families as well as substantial social and economic costs to the society. Early rehabilitation is highly important for restoring lost skills and functioning, but often very difficult given the severity and extent of the TBI symptoms and the high strain that the available rehabilitation methods put on the patients. Music therapy is a highly motivating, versatile, and applicable form of TBI rehabilitation, but currently there is little scientific evidence for its efficacy or mechanisms in the TBI population. The purpose of the present project is to determine the long-term effect of Music-based Neurological Rehabilitation (MBNR) on cognitive, motor, emotional, and social recovery after TBI in adolescents and young adults, and to study the neural mechanisms that underlie behavioural recovery and the efficacy of music.

The study is a single-blind, cross-over randomized controlled trial (RCT) involving 60 adolescents and young adults with a subacute moderate / severe TBI. During an 18-month follow-up, the patients receive MBNR (30 session, 3 x week, 1 hour sessions) and/or Standard Care (SC). The MBNR intervention utilizes structured cognitive-motor training with drums and creative musical expression (music playing, song writing) with piano that are geared towards engaging and training attention, executive functions, working memory, and upper-extremity functions and for enhancing emotional self-expression, adjustment, and mood after TBI. The SC consists of other types of conventional rehabilitation (e.g., physical therapy, neuropsychological rehabilitation) and medical care for TBI provided in private or public health care. Half of the patients receive the MBNR intervention during the first 10-week period and half during the second 10-week period (in addition, all patients receive SC during the whole follow-up period).

Outcome measures comprise neuropsychological tests (measuring executive functions, attention, reasoning, and working memory and learning), neurological scales (measuring neurological symptoms, functional outcome, adjustment, and participation), motor tests (measuring motor dexterity, coordination, and upper limb functioning), and structural and functional magnetic resonance imaging (MRI/fMRI, measuring gray and white matter structure and integrity and auditory-motor neural processing) performed at the start of the study (baseline), after the first 10-week period (3-month stage) and after the second 10-week period (6-month stage). At these time points as well as 12 months later (18-month stage), the patients and their caregivers are also given questionnaires measuring executive functions, depression symptoms, quality of life, and caregiver well-being and burden.

ELIGIBILITY:
Inclusion Criteria:

* moderate-severe TBI that has occurred ≤ 24 months ago
* cognitive symptoms
* right-handed
* living in the Helsinki metropolitan area
* able to understand the purpose of the study and provide informed consent

Exclusion Criteria:

* prior neurological or psychiatric illness or substance abuse
* prior auditory deficits (severe hearing loss, tinnitus, etc.)
* contraindications for MRI (pacemaker, metal prosthesis, etc.)

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Executive Functions during an 18-month follow-up | Baseline, 3 months, 6 months, and 18 months
  Executive Functions (EF) are assessed using the Behavior Rating Inventory of Executive Functions (BRIEF-A, both self-report and informant-report versions) questionnaire and following cognitive tests: Frontal Assessment Battery (FAB, measure of overall EF), Number-Letter Task (measure of set-shifting ability), Simon Task (measure of inhibition), and Auditory N-back Task (measure of working memory updating). The cognitive tests are performed at the baseline, 3-month, and 6-month stages and the BRIEF-A is performed at the baseline, 3-month, 6-month, and 18-month stages. Changes from baseline to each follow-up point (3-month / 6-month / 18-month) and between the follow-up points are evaluated.
Change in Focused and Sustained Attention during a 6-month follow-up | Baseline, 3 months, and 6 months
  Focused and Sustained Attention is assessed using the Sustained Attention to Response Task (SART) performed at the baseline, 3-month, and 6-month stages. Changes from baseline to each follow-up point (3-month / 6-month) and between the follow-up points are evaluated.
Change in Verbal Working Memory and Learning during a 6-month follow-up | Baseline, 3 months, and 6 months
  Verbal Working Memory and Learning are assessed using the Digit Span subtest of the Wechsler Adult Intelligence Scale IV (WAIS-IV) and the Word List I & II subtests of the Wechsler Memory Scale III (WMS-III) performed at the baseline, 3-month, and 6-month stages. Changes from baseline to each follow-up point (3-month / 6-month) and between the follow-up points are evaluated.
Change in Verbal and Non-Verbal Reasoning during a 6-month follow-up | Baseline, 3 months, and 6 months
  Verbal and Non-Verbal Reasoning are assessed using the Similarities and Block Design subtests of the Wechsler Adult Intelligence Scale IV (WAIS-IV) performed at the baseline, 3-month, and 6-month stages. Changes from baseline to each follow-up point (3-month / 6-month) and between the follow-up points are evaluated.

SECONDARY OUTCOMES:
Change in Upper-Extremity Motor Functions during a 6-month follow-up | Baseline, 3 months, and 6 months
  Upper-Extremity Motor Functions are assessed using the Purdue Pegboard Test (PPT, measure of fine and gross motor dexterity and coordination), the Action Research Arm Test (ARAT, measure of fine and gross upper limb functioning), and the Box and Block Test (BBT, measure of unilateral manual dexterity) performed at the baseline, 3-month, and 6-month stages. Changes from baseline to each follow-up point (3-month / 6-month) and between follow-up points are evaluated.
Change in Depression during an 18-month follow-up | Baseline, 3 months, 6 months, and 18 months
  Depression is assessed using the Beck Depression Inventory II (BDI-II, self-report version) questionnaire performed at the baseline, 3-month, 6-month, and 18-month stages. Changes from baseline to each follow-up point (3-month / 6-month / 18-month) and between the follow-up points are evaluated.
Change in Quality of Life during an 18-month follow-up | Baseline, 3 months, 6 months, and 18 months
  Quality of Life is assessed using the Quality of Life after Brain Injury (QOLIBRI, both self-report and informant-report versions) questionnaire performed at the baseline, 3-month, 6-month, and 18-month stages. Changes from baseline to each follow-up point (3-month / 6-month / 18-month) and between the follow-up points are evaluated.
Change in Emotional Well-being of Family Members during an 18-month follow-up | Baseline, 3 months, 6 months, and 18 months
  Emotional Well-being of Family Members is assessed using the General Health Questionnaire (GHQ) and the Modified Caregiver Appraisal Scale (MPAI) given to the family member of the patient at the baseline, 3-month, 6-month, and 18-month stages. Changes from baseline to each follow-up point (3-month / 6-month / 18-month) and between the follow-up points are evaluated.
Change in Structural and Functional Neuroplasticity during a 6-month follow-up | Baseline, 3 months, and 6 months
  Structural and Functional Neuroplasticity is measured using structural and functional magnetic resonance imaging (MRI/fMRI) scanning performed at the baseline, 3-month, and 6-month stages. Overall, the purpose of the MRI/fMRI is to determine the exact location and size of the lesions and other pathological changes caused by the TBI and to study the changes in grey matter volume (using voxel-based morphometry, VBM), white matter volume and organization (using diffusion tensor imaging, DTI), and auditory-motor activity and connectivity (using fMRI) that take place in different brain areas during the 6-month follow-up and to correlate these changes to behavioral recovery. Changes from baseline to each follow-up point (3-month / 6-month) and between the follow-up points are studied.

CONTACTS AND LOCATIONS:
Overall Officials: Teppo Sarkamo, PhD, Principal Investigator — University of Helsinki; Mari Tervaniemi, PhD, Study Director — University of Helsinki; Anne Vehmas, MD, Study Chair — Kapyla Rehabilitation Centre, Helsinki, Finland
Locations (3):
- Finland (3):
  - Helsinki University Central Hospital / Brain Injury Outpatients Clinic, Helsinki
  - Validia Rehabilitation Helsinki, Helsinki
  - Lohja Hospital, Department of Neurology, Lohja

REFERENCES:
- [Derived] Sihvonen AJ, Siponkoski ST, Martinez-Molina N, Laitinen S, Holma M, Ahlfors M, Kuusela L, Pekkola J, Koskinen S, Sarkamo T. Neurological Music Therapy Rebuilds Structural Connectome after Traumatic Brain Injury: Secondary Analysis from a Randomized Controlled Trial. J Clin Med. 2022 Apr 14;11(8):2184. doi: 10.3390/jcm11082184. PMID 35456277
- See also: Cognitive Brain Research Unit, Helsinki University — http://www.cbru.helsinki.fi/
- See also: Finnish Centre of Excellence in Interdisciplinary Music Research, University of Jyvaskyla — https://www.jyu.fi/hum/laitokset/musiikki/en/research/coe
- See also: Validia Rehabilitation Helsinki — http://www.validia.fi/
- See also: Cognition and Brain Plasticity Group, University of Barcelona — http://www.brainvitge.org/index.php